CLINICAL TRIAL: NCT03693235
Title: Adequate Bending Angle of a Lightwand for Tracheal Intubation
Brief Title: Adequate Bending Angle of a Lightwand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30-2018-44
Record Dates: First submitted 2018-09-30; First posted 2018-10-02 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Tracheal Intubation
Keywords: Tracheal Intubation; Lightwand

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 70 degrees (Experimental): During tracheal intubation using a lightwand, the tracheal tube combined with a lightwand will be bent by 70 degrees.
  Interventions: Procedure: bending angle of a lightwand
- 80 degrees (Experimental): During tracheal intubation using a lightwand, the tracheal tube combined with a lightwand will be bent by 80 degrees.
  Interventions: Procedure: bending angle of a lightwand
- 90 degrees (Experimental): During tracheal intubation using a lightwand, the tracheal tube combined with a lightwand will be bent by 90 degrees.
  Interventions: Procedure: bending angle of a lightwand

INTERVENTIONS:
Procedure: bending angle of a lightwand — For tracheal intubation, investigators will bend the tracheal tube combined a lightwand by assigned angles (70, 80, or 90 degrees) for each patient. Next a practitioner will perform tracheal intubation with the bent tube.

SUMMARY:
For tracheal intubation with a lightwand, adequate bending angle was not exactly investigated. The purpose of the study is compare three bending angles of lightwands for safe and efficient tracheal intubation.

DETAILED DESCRIPTION:
Lightwands are very useful device for difficult airway management due to small moth opening, weak teeth, and cervical spine instability. Experienced clinicians use a lightwand while bending it adequately. However, there has been not previous studies to investigate the adequate angle to bend it.

This randomized controlled trial is to compare three angles (70, 80, and 90 degrees) as bending angle of lightwands for safe and efficient tracheal intubation in cases which require the use of lightwands.

ELIGIBILITY:
Inclusion Criteria:

* patients who require use of a lightwand for tracheal tubes (i.e. small mouth opening, weak teeth, cervical spine instability)

Exclusion Criteria:

* patients who refuse to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
sore throat | After surgery
  After surgery, investigators evaluate VAS score for sore throat of the patients.
Intubation time | Intraoperative
  from initiation of tracheal intubation with a lightwand after bending it to completion of tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D., PhD., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Agro F, Hung OR, Cataldo R, Carassiti M, Gherardi S. Lightwand intubation using the Trachlight: a brief review of current knowledge. Can J Anaesth. 2001 Jun;48(6):592-9. doi: 10.1007/BF03016838. PMID 11444456
- [Background] Chen J, Luo W, Wang E, Lu K. Optimal bent length of lightwand for intubation in adults: a randomized, prospective, comparative study. J Int Med Res. 2012;40(4):1519-31. doi: 10.1177/147323001204000432. PMID 22971505
- [Background] Davis L, Cook-Sather SD, Schreiner MS. Lighted stylet tracheal intubation: a review. Anesth Analg. 2000 Mar;90(3):745-56. doi: 10.1097/00000539-200003000-00044. No abstract available. PMID 10702469
- [Background] Kim J, Im KS, Lee JM, Ro J, Yoo KY, Kim JB. Relevance of radiological and clinical measurements in predicting difficult intubation using light wand (Surch-lite) in adult patients. J Int Med Res. 2016 Feb;44(1):136-46. doi: 10.1177/0300060515594193. Epub 2015 Dec 7. PMID 26647074
- [Background] Szigeti CL, Baeuerle JJ, Mongan PD. Arytenoid dislocation with lighted stylet intubation: case report and retrospective review. Anesth Analg. 1994 Jan;78(1):185-6. doi: 10.1213/00000539-199401000-00034. No abstract available. PMID 8267162
- [Derived] Won D, Lee JM, Lee J, Hwang JY, Kim TK, Chang JE, Kim H, Ma S, Min SW. A pilot study comparing three bend angles for lighted stylet intubation. BMC Anesthesiol. 2021 May 17;21(1):148. doi: 10.1186/s12871-021-01369-8. PMID 34000987